CLINICAL TRIAL: NCT06155734
Title: Fluorescence Guided Minimally-Invasive Resection Of Abdominal Paragangliomas Using Indocyanine Green
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Alexander Vahrmeijer, Principle investigator, oncologic surgeon, MD, PhD, Leiden University Medical Center
Other Study IDs: nWMO_GLL_1
Record Dates: First submitted 2023-11-16; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Paraganglioma
Keywords: Fluorescence Guided Surgery
MeSH Terms: conditions — Paraganglioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retrospective intervention cohort
  Interventions: Drug: Fluorescence guided identification using indocyanine green

INTERVENTIONS:
Drug: Fluorescence guided identification using indocyanine green — During minimally invasive surgery using intravenous administration of indocyanine green (ICG) near-infrared fluorescence imaging will be applied to identify and treat paragangliomas

SUMMARY:
This study is exploring whether it's possible to detect paragangliomas (a rare type of tumor) during minimally invasive surgery by using a technique called near-infrared fluorescence imaging, guided by a substance called indocyanine green (ICG). The goal is to see if this method can help surgeons identify and treat paragangliomas more accurately and during minimally invasive procedures.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with abdominal paraganglioma and underwent minimally-invasive surgical resection

Exclusion Criteria:

* Open surgical procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients >18yo diagnosed with abdominal paragangliomas which underwent surgical resection
Sampling Method: Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
Feasibility of real-time in-vivo identification of suspected paraganglioma's using Near-Infrared-fluorescence ICG imaging | perioperatively/periprocedurally, within 30 minutes after intravenous administration of the fluorescent dye, up until a maximum of 120 minutes after start of surgery.
  The primary outcome of this retrospective study is the ability to visually detect the proportion (%) of suspected pre-operatively identified lesions (paraganglioma) in the abdomen during minimally invasive procedures using Near-Infrared-fluorescence ICG imaging

SECONDARY OUTCOMES:
Accuracy of the detection of suspected lesions using Near-Infrared-fluorescence ICG imaging | Postoperatively, at the moment the definitive pathology result is known, approximately five days after surgery
  The secondary outcome of this retrospective study is the accuracy, measured by sensitivity and specificity to identify abdominal paragangliomas using using Near-Infrared-fluorescence ICG imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided